CLINICAL TRIAL: NCT01229696
Title: Continuous Popliteal Nerve Blocks: Effect of Perineural Catheter Tip Location Relative to the Sciatic Nerve Bifurcation on Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Popliteal Bifurcation
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Popliteal Nerve Block; Foot Surgery; Ankle Surgery; Popliteal Bifurcation
Keywords: Popliteal; UCSD; Postoperative pain; Foot surgery; Ankle surgery; Popliteal Catheter; Popliteal Nerve Block; Lower extremity surgery; Bifurcation; Catheter Insertion Site
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- At Bifurcation (Active Comparator): Patients randomized to this group will receive a sciatic nerve block placed at the bifurcaton of the sciatic nerve and outcome measures will be tested.
  Interventions: Procedure: Catheter Placed At Bifurcation
- 5cm Above Bifurcation (Active Comparator): Patients randomized to this group will receive a sciatic nerve block placed 5cm above the bifurcaton of the sciatic nerve and outcome measures will be tested.
  Interventions: Procedure: Catheter Placed 5cm Above Bifurcation

INTERVENTIONS:
Procedure: Catheter Placed At Bifurcation — Patients randomized to this group will receive a sciatic nerve block placed at the bifurcaton of the sciatic nerve and outcome measures will be tested.
  Arms: At Bifurcation
Procedure: Catheter Placed 5cm Above Bifurcation — Patients randomized to this group will receive a sciatic nerve block placed 5cm above the bifurcaton of the sciatic nerve and outcome measures will be tested.
  Arms: 5cm Above Bifurcation

SUMMARY:
Research study to determine the relationship between perineural catheter tip location relative to the sciatic nerve bifurcation and postoperative analgesia for continuous popliteal nerve blocks.

DETAILED DESCRIPTION:
Hypothesis: During a continuous popliteal nerve block, postoperative analgesia will be improved with the perineural catheter tip at the level of the sciatic nerve bifurcation compared to when the catheter tip is 5 cm cephalad/proximal to the bifurcation.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery with a popliteal perineural catheter for postoperative analgesia
* age 18 years or older

Exclusion Criteria:

* pregnancy
* inability to communicate with the investigators and hospital staff
* incarceration
* clinical neuropathy in the surgical extremity
* chronic high-dose opioid use
* a history of opioid abuse
* surgery outside of ipsilateral sciatic and saphenous nerve distributions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Average Pain | 1 Day following surgery
  The average pain in the three hours previous to a phone call the day following surgery as measured on a numeric rating scale (0-10, 0=no pain, 10=worst imaginable pain).

SECONDARY OUTCOMES:
Analgesic Use | 1 day following surgery
  Total oral opioid use since surgery and total IV analgesics if any.
Sleep Disturbances | 1 day following surgery
  Total number of times patient woke due to pain the night following surgery.
Infusion Side Effects | 1 day following surgery
  Numbness of foot and toes on a 0-10 scale where 0=no numbness and 10=complete numbness.
Satisfaction of pain control | 1 day following surgery
  Patients will give an answer on a 0-10 scale where 0=completely unsatisfied wiht pain control and 10=completely satisfied with pain control.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Centers (Hillcrest and Thornton), San Diego, California, United States